CLINICAL TRIAL: NCT06534749
Title: Ultrasound Screening of Congenital Anomalies of Kidney and Urinary Tract in Neonates
Acronym: CAKUT
Status: Active, not recruiting | Type: Observational
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Sara Mabrouk Elghoul, lectrurer of pediatric nephrology, Tanta University
Other Study IDs: 36264PR377/10/23
Record Dates: First submitted 2024-07-30; First posted 2024-08-02 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Urinary Tract Anomalies; Kidney; Anomaly
MeSH Terms: conditions — Congenital Abnormalities | interventions — Ultrasonography

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ultrasound — Ultrasound screening: by (SonoScape A6, Yizhe Building, Yuquan, Road Shenzhen, 518051, China). General-purpose diagnostic abdominal ultrasound equipment was used, with a 7.5-MHz linear-type probe. Screenings will be performed by radiologist with appropriate practice. The ultrasound examination will take 10 min for each patient. The recordings will consist of two bilateral renal images will be obtained and one transverse and longitudinal images. The urinary bladder will be observed with the patient in a supine position, and images will be recorded when abnormalities will be identified. The following will be investigated by ultrasound: number, size (including differences between sides), and location of the kidneys; pelvic dilatation; echogenicity, and other findings indicating cysts or tumours. Shape and wall thickening of the urinary bladder, as well as ureter dilatation, will be also examined

SUMMARY:
This cross sectional study will be conducted to investigate the incidence of the congenital anomalies of kidney and urinary tracts in neonates born or admitted at Tanta University Hospital.

DETAILED DESCRIPTION:
This cross sectional study will be conducted for one year from October 2023 to October 2024 at Pediatric and Radiology Departments Tanta University Hospital (TUH).

This study will be conducted on neonates who will be born or admitted at Tanta University Hospital.

All patients included in the study will be subjected to: history taking, clinical examination and Ultrasound screening: by (SonoScape A6, Yizhe Building, Yuquan, Road Shenzhen, 518051, China). General-purpose diagnostic abdominal ultrasound equipment was used, with a 7.5-MHz linear-type probe. Screenings will be performed by radiologist with appropriate practice. The ultrasound examination will take 10 min for each patient. The recordings will consist of two bilateral renal images will be obtained and one transverse and longitudinal images. The urinary bladder will be observed with the patient in a supine position, and images will be recorded when abnormalities will be identified. The following will be investigated by ultrasound: number, size (including differences between sides), and location of the kidneys; pelvic dilatation; echogenicity, and other findings indicating cysts or tumours. Shape and wall thickening of the urinary bladder, as well as ureter dilatation, will be also examined.

ELIGIBILITY:
Inclusion Criteria:

* Neonates in the first month of life.

Exclusion Criteria:

* no exclusions

Ages: 3 Days to 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: neonates who will be born or admitted at Tanta University Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2023-10-28 (Actual); Primary Completion 2024-10 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Incidence of CAKUT in neonates | one year
  investigate the incidence of the congenital anomalies of kidney and urinary tracts in neonates born or admitted at Tanta University Hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Sara Mabrouk Mohamed Elghoul, MD, Principal Investigator — Tanta University
Locations (1):
- Sara Mabrouk Mohamed Elghoul, Tanta, Tanta, Qism 1, Egypt

IPD SHARING:
Plan to Share IPD: Undecided